CLINICAL TRIAL: NCT05670574
Title: Surgery With Extended (D3) Mesenterectomy for Small Bowel Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Helse Sor-Ost (Other Government); University of Geneva, Switzerland (Other); Oslo University Hospital (Other); CarciNor (Unknown)
Responsible Party: Principal Investigator, Dejan Ignjatovic, Professor, University Hospital, Akershus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1286
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Small Bowel Cancer; Small Bowel Carcinoid Tumor; Quality of Life; Lymph Node Metastases; Tumor Metastasis
Keywords: Small bowel cancer; Extended mesenterectomy; Lymph node metastases; Tumor feeding vessel; Quality of life
MeSH Terms: conditions — Lymphatic Metastasis; Neoplasm Metastasis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Testing three new surgical techniques for small bowel tumors. Tumor feeding vessel and vascular anatomy of each patients is identified preoperatively on CT scan and based on this we produce a 3D reconstruction. Based on tumor location we choose one of the three techniques and perform extended D3 mesenterectomy. The results will be reported on as described in the "project description" section
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery with extended (D3) mesenterectomy for small bowel tumors

SUMMARY:
The study is designed to investigate the safety and efficacy of central D3 lymphadenectomy in cases of small bowel tumors. Such dissection is under debate; consensus guidelines are vague when it comes to surgical techniques and practice is highly variable.

DETAILED DESCRIPTION:
Cancer of the small intestine is rare. Consensus practice on surgical technique have been difficult to reach, both on lymph node dissection level and on strategic choices according to tumor localization and -type. Evidence is strong for systematic and radical lymphadenectomy for neuroendocrine tumors (NET) and adenocarcinomas. This study includes a series of prospective and consecutive patients operated with central (D3) lymphadenectomy. Key points are preoperative mapping of vascular anatomy to facilitate personalized surgery with radical lymphadenectomy to the mesenterial root, both anterior and posterior to the superior mesenteric vessels. Three different surgical techniques (plus one subgroup) are used, and will be reported on, according to tumor localization and -type. Complications, perioperative morbidity and mortality, operating time and length of hospital stay will be noted, as well as tumor types, number of tumors, mesenteric mass size, resection types and margins, and the anatomical distribution of tumors. Patient outcome during 2- and 5-year follow up will be reported. We will investigate the accuracy of the preoperative vascular anatomy reconstructions and eventual procedure-specific complications. Still, the main outcome measures are the lymph node yield: number of lymph nodes gained in the D2 and D3 areas.

Patients are included in the study "Safe extended (D3) mesenterectomy for small bowel tumors" - REK number 19898. Patients are given an informed consent formula. Inclusion criteria are patients with small bowel tumor(s) of probable or confirmed neoplastic nature capable of consent and without general inoperability properties. The ENETS Neuroendocrine Tumor Centre of Excellence at Oslo University Hospital approves and recommends surgery for patients with NET. All patients shall have their mesenterial vascular anatomy reconstructed in 3D preoperatively, for both arteries and veins. The reconstruction is made by manual segmentation based on biphasic CT scans of their abdomens.

The surgical-oncological aim is the same for both open and minimally invasive access surgery: an intact and continuous specimen with tumor and mesentery in one piece including unbroken and correct anatomical tissue planes. We define the D3 volume to include all lipolymphatic tissue anterior and posterior to the superior mesenteric vessels limited by arterial and venous branches to and from the tumor-bearing segment of bowel. Dissection is made along the blood vessels cranially and caudally. Mesenteric nodal masses and fibrosis and desmoplasia are carefully dissected from the underlying blood vessels to be saved by exposing and dividing the vessel sheets

ELIGIBILITY:
Inclusion Criteria:

* Patients included must be able to fill in an informed, written consent and to understand its implications and contents and to participate in the follow-up
* Radiologically/scintigraphically/histologically verified extraduodenal tumor(-s) in the small bowel and/or in the mesentery of the small bowel
* No signs of inoperability
* Fit for general anesthetics

Exclusion Criteria:

* Extraduodenal small bowel tumors verified as GIST or benign tumor
* Widespread lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of lymph nodes in total in D2 and D3 areas | 1 month
Number of positive lymph nodes in D2 and D3 areas | 1 month

SECONDARY OUTCOMES:
Complications | 30 days
Peroperative blood loss | 30 days
Hospitalization time | 1-90 days
Operation time | Intraoperative
Tumor type | 30 days
Presence and size of mesenteric mass | 30 days
Resection type and -margins | 30 days
30-day mortality | 30 days
2-year follow-up | 2 years
5-year follow-up | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Ignjatovic, MD PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lorenskog, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vasic T, Stimec M, Stimec BV, Edwin B, Ignjatovic D. Lymphatic and vascular anatomy define surgical principles for radical treatment of distal duodenal and proximal jejunal tumors. Surg Endosc. 2025 Aug;39(8):5421-5429. doi: 10.1007/s00464-025-11909-9. Epub 2025 Jul 7. PMID 40624418
- [Derived] Vasic T, Stimec MB, Stimec BV, Kjaestad E, Ignjatovic D. Jejunal Lymphatic and Vascular Anatomy Defines Surgical Principles for Treatment of Jejunal Tumors. Dis Colon Rectum. 2025 May 1;68(5):553-561. doi: 10.1097/DCR.0000000000003644. Epub 2025 Feb 12. PMID 39936801